CLINICAL TRIAL: NCT07374913
Title: Study of the Familial Phenotype Associated With Mutations in the COL4A1 and COL4A2 Genes
Brief Title: COL4A1COL4A2: Study of Pathological Conditions Involving Multiple Organs Caused by Mutations in the COL4A1 and COL4A2 Genes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Simona Balestrini, Clinical Professor, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COL4A1COL4A2
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: COL4A1\2; COL4A1-Related Brain Small Vessel Disease With Haemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COL4A1/2 variant carriers (Experimental): This is a single-arm observational study with defined participant subgroups. No experimental interventions are administered.
  Participants include individuals with pathogenic or likely pathogenic COL4A1 or COL4A2 variants and their first-degree family members. All participants undergo observational data collection through a structured clinical questionnaire. Adult family members who are confirmed or suspected carriers of the mutation are additionally offered non-invasive diagnostic assessments, including ophthalmological examinations (anterior segment photography and optical coherence tomography) and cardiological evaluations (resting ECG, ambulatory ECG, and echocardiography), performed as part of routine clinical care.
  A blood sample is collected from affected individuals and adult non-carrier relatives for exploratory laboratory analyses of matrix metalloproteinase (MMP2/MMP9) activity. Non-carrier relatives serve as a biological control group for these analyses.
  Interventions: Diagnostic Test: Ophtalmological and cardiological screening

INTERVENTIONS:
Diagnostic Test: Ophtalmological and cardiological screening — Participants who are confirmed or suspected carriers of a COL4A1 or COL4A2 pathogenic variant are offered non-invasive diagnostic ophthalmological and cardiological screening to assess potential organ involvement associated with the genetic condition.
  The ophthalmological screening includes anterior segment photography of both eyes and optical coherence tomography (OCT) to evaluate retinal structure, macular thickness, and retinal nerve fiber layer.
  The cardiological screening includes a resting electrocardiogram (ECG), ambulatory ECG monitoring, and transthoracic echocardiography to assess heart rhythm, conduction, and cardiac structure and function.
  These procedures are performed within routine clinical care settings and are used solely for observational and diagnostic purposes; no therapeutic intervention is administered as part of the study.

SUMMARY:
This observational and diagnostic study aims to better understand the clinical features and biological mechanisms associated with mutations in the COL4A1 and COL4A2 genes, which are known to cause a rare inherited small-vessel disease affecting the brain and other organs. These mutations can lead to a wide range of symptoms involving the brain, eyes, heart, blood vessels, kidneys, and muscles, and affected individuals within the same family may show very different clinical manifestations.

The study will systematically collect clinical and diagnostic information from individuals with confirmed COL4A1/COL4A2 mutations and their first-degree family members, including both affected and unaffected relatives. Family members who carry, or may carry, the mutation will be offered non-invasive eye and heart examinations to detect early or previously unrecognized organ involvement.

In addition, blood samples will be analyzed to study the activity of specific enzymes called matrix metalloproteinases (MMP2 and MMP9), which are thought to play a role in blood vessel damage in this condition. By linking genetic findings, clinical features, and laboratory data, the study seeks to clarify how these mutations cause disease and to identify early signs of organ involvement.

The overall goal of the study is to improve early diagnosis, guide the development of routine multi-organ screening strategies for affected individuals and families, and support future research toward targeted treatments.

DETAILED DESCRIPTION:
This is an observational, prospective cohort study designed to characterize the clinical spectrum and underlying biological mechanisms associated with pathogenic or likely pathogenic variants in the COL4A1 and COL4A2 genes. These genes encode type IV collagen, a key structural component of basement membranes, and their alteration is associated with a rare autosomal dominant small-vessel disease with variable multi-organ involvement.

Individuals with a confirmed COL4A1/COL4A2 mutation identified through clinical genetic testing will be invited to participate together with their first-degree family members. Adult relatives who are confirmed carriers or are suspected carriers of the same mutation will be included in the diagnostic component of the study. Adult non-carrier relatives will serve as controls for selected laboratory analyses.

Participants will complete a structured questionnaire collecting standardized information on neurological, ophthalmological, cardiovascular, renal, muscular, and other systemic manifestations. Carrier or suspected carrier relatives will be offered non-invasive diagnostic screening, including ophthalmological assessments (anterior segment photography and optical coherence tomography) and cardiological evaluations (resting electrocardiogram, ambulatory ECG monitoring, and echocardiography), performed within routine clinical care settings.

A blood sample will be collected from affected individuals and adult non-carrier relatives. Plasma will be stored and analyzed to assess the activity of matrix metalloproteinases MMP2 and MMP9 using established laboratory techniques. These analyses aim to explore molecular pathways potentially involved in vascular and tissue damage associated with COL4A1/COL4A2 variants.

The study does not include a scheduled follow-up; data are collected at a single time point per participant. Results will be analyzed using descriptive and exploratory statistical methods to evaluate the prevalence and pattern of multi-organ involvement and to explore associations between genetic variants, clinical features, and laboratory findings.

The knowledge gained from this study is intended to support improved clinical characterization of COL4A1/COL4A2-related disease, inform the development of structured multi-organ screening strategies, and provide a foundation for future therapeutic research

ELIGIBILITY:
Inclusion Criteria:

* Individuals (pediatric or adult) with a pathogenic or likely pathogenic mutation in the COL4A1 or COL4A2 genes and a clinical phenotype consistent with small vessel disease.
* Adult first-degree family members (parents, siblings, or children) who are confirmed carriers or suspected carriers of the same COL4A1/COL4A2 mutation.
* Adult first-degree family members who are non-carriers of the pathogenic mutation and who agree to provide a blood sample to be used as controls for laboratory analyses.
* Ability to provide written informed consent; for minors, consent provided by a parent or legal guardian.

Exclusion Criteria:

* Refusal or inability to provide informed consent.
* Individuals who do not meet the inclusion criteria above.
* Any condition that, in the opinion of the investigators, would preclude participation in study procedures or reliable data collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence and pattern of multi-organ involvement | Single time point at study enrollment (baseline assessment)

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCSS, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No